CLINICAL TRIAL: NCT01569607
Title: Structurally Reorganizing Motor Cortex in Stroke Patients Through Hebbian-type Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathrin Buetefisch (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Cathrin Buetefisch, Dr. Cathrin Buetefisch, MD, PhD, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00052053; R21HD067906-01A1 (NIH); SRMC21 (Other: Other)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Stroke
Keywords: Neurophysiology; Transcranial Magnetic Stimulation (TMS); Neurology; Stroke; Physical Medicine and Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hebbian-type Stimulation (Experimental): Participants will be randomized to receive motor training with Hebbian-type stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham Stimulation (Sham Comparator): Participants will be randomized to receive sham stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Training sessions for 5 days in a row
  Arms: Hebbian-type Stimulation
Device: Sham stimulation — Sham stimulation
  Arms: Sham Stimulation

SUMMARY:
Stroke is a leading cause of morbidity in the United States but identification of treatment strategies to improve outcome is limited by the incomplete understanding of the mechanisms of recovery. Motor cortex (M1) reorganization plays a major-role in the recovery of motor deficits post-stroke; hence the importance for further development of rehabilitative strategies that utilize this potential for recovery.

In Specific Aim 1, investigators will determine if repeated exposure to training combined with Hebbian-type M1 stimulation enhances functional M1 reorganization in lesioned M1 of stroke patients.

In Specific Aim 2, investigators will determine if repeated exposure to training combined with Hebbian-type M1 stimulation enhances structural cortical reorganization in lesioned M1 of stroke patients and to explore whether these structural changes are related to the training induced functional cortical reorganization.

The overall goal of this project is to determine the effect of Hebbian- type stimulation on both, functional and structural brain reorganization, thereby obtaining indirect evidence for the neuronal substrate underlying training related improvement and maintenance of motor function in stroke patients. This knowledge may have a substantial positive impact on treatment for stroke patients that may significantly improve recovery and could move the field of neuro-rehabilitation forward.

DETAILED DESCRIPTION:
Stroke is a leading cause of morbidity in the United States but identification of treatment strategies to improve outcome is limited by the incomplete understanding of the mechanisms of recovery. Motor cortex (M1) reorganization plays a major-role in the recovery of motor deficits post-stroke; hence the importance for further development of rehabilitative strategies that utilize this potential for recovery. Non-invasive cortical stimulation can enhance the beneficial effects of motor training on performance and functional plasticity of motor cortex. Among the different approaches used in these studies, Hebbian-type M1 stimulation is particularly intriguing, as it seems to be more effective when compared to random M1 stimulation. There is emerging evidence that motor training or cortical stimulation related improvement of function are associated with increases in the grey matter of targeted brain areas. While there is therefore some evidence supporting structural reorganization in human M1 in response to motor learning and cortical stimulation, the mechanisms underlying these changes and their relationship to functional plasticity are not known. A better understanding of the sequences of events is critical to development of optimal therapeutic interventions to improve recovery following stroke.

In Specific Aim 1, investigators will determine if repeated exposure to training combined with Hebbian-type M1 stimulation enhances functional M1 reorganization in lesioned M1 of stroke patients.

In Specific Aim 2, investigators will determine if repeated exposure to training combined with Hebbian-type M1 stimulation enhances structural cortical reorganization in lesioned M1 of stroke patients and to explore whether these structural changes are related to the training induced functional cortical reorganization.

The overall goal of this project is to determine the effect of Hebbian- type stimulation on both, functional and structural brain reorganization, thereby obtaining indirect evidence for the neuronal substrate underlying training related improvement and maintenance of motor function in stroke patients. This knowledge may have a substantial positive impact on treatment for stroke patients that may significantly improve recovery and could move the field of neuro-rehabilitation forward.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Single cerebral ischemic infarction > 6 month affecting the primary motor output system of the hand at a cortical (M1) level as defined by MRI of the brain
* At the time of cerebral infarct a motor deficit of hand of MRC of <4- of wrist and finger extension/flexion movement
* Good recovery of hand function as defined by MRC of 4 or 4+ of wrist- and finger extension/flexion movements
* Ability to perform wrist extension movements
* No other neurological disorder
* No intake of CNS active drugs
* Ability to give informed consent
* Ability to meet criteria of inclusion experiment
* No major cognitive impairment
* No contraindication to TMS or MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Buetefisch, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Revill KP, Haut MW, Belagaje SR, Nahab F, Drake D, Buetefisch CM. Hebbian-Type Primary Motor Cortex Stimulation: A Potential Treatment of Impaired Hand Function in Chronic Stroke Patients. Neurorehabil Neural Repair. 2020 Feb;34(2):159-171. doi: 10.1177/1545968319899911. Epub 2020 Jan 24. PMID 31976804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between March 2012 and August 2016.
Pre-assignment Details: Participants completed the eligibility phase prior to being randomized to a study arm. Of the 48 participants that provided consent, 22 were eligible for participation and were randomized to an intervention.
Groups:
- Hebbian-type Stimulation: Participants were randomized to receive motor training with Hebbian-type stimulation.
  Repetitive Transcranial Magnetic Stimulation (rTMS): Training sessions for 5 days in a row
- Sham Stimulation: Participants were randomized to receive sham stimulation.
  Sham stimulation: Sham stimulation
Period: Overall Study
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants that were randomized to a study arm and received an intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hebbian-type Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Primary Motor Cortex (M1) Excitability Derived From Stimulus Response Curve
Description: Motor evoked potential (MEP) amplitudes were measured prior to treatment (baseline), one week after the treatment (post-training 1), and 4 weeks after treatment (post-training 2).The MEP is elicited by transcranial magnetic stimulation (TMS) at increased intensity. Its amplitude is measured from peak to peak and expressed in millivolts (mV). Measured MEP amplitudes were plotted against the intensity to create a stimulus response curve (SRC). Long-lasting increases in MEP amplitude indicate increases in motor cortex excitability and are associated with motor learning.
Time Frame: Baseline, Post-Training 1 (1 Week), Post-Training 2 (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
millivolts
  Baseline | 4.68 (5.65) | 9.09 (11.28)
  Post-Training Week 1 | 5.01 (5.96) | 8.04 (9.28)
  Post-Training Week 4 | 2.66 (2.55) | 7.66 (10.67)

2. Secondary Outcome: Mean Time to Completion for Jebsen Hand Function Test (JTT)
Description: The JTT provides a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living assessing the speed of performance. Total score is the sum of time taken for each sub-test, which were normalized to standard scores (also expressed in seconds).Total scores range from +1 to -1 where -1 indicates best function.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | .38 (.23) | .49 (.21)
  Post-Training Week 1 | .34 (.26) | .45 (.20)
  Post-Training Week 4 | .31 (.26) | .44 (.21)

3. Secondary Outcome: Mean Peak Acceleration of Wrist Extension Movements
Description: Mean peak acceleration was measured at baseline, one week after the treatment (post-training 1), and four weeks after the treatment (post-training 2). Increases in the mean peak acceleration of the trained wrist extension movements indicate motor learning. Acceleration was measured in g; a symbol for the average acceleration produced by gravity at the Earth's surface.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Three participants from both arms were removed from the data analysis due to errors in data collection yielding uninterpretable results.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 7 | 7
g
  Baseline | .61 (.48) | .60 (.32)
  Post-Training Week 1 | .72 (.32) | .79 (.49)
  Post-Training Week 4 | .71 (.32) | .81 (.47)

4. Secondary Outcome: Mean Reaction Time of Wrist Extension Movements
Description: Subjects will be asked to perform 7 auditory-cued ballistic wrist extensions before and after motor training. Electromyographic (EMG) activity recorded during the ballistic wrist extensions will be used to measure reaction time. Reaction time is the length of time between the auditory cue and the onset of the movement-related EMG burst of the extensor carpi ulnaris muscle. A longer time indicated longer time to reaction.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 7 | 7
milliseconds
  Baseline | 238.1 (77.40) | 257.14 (88.13)
  Post-Training Week 1 | 238.43 (36.38) | 224.59 (63.69)
  Post-Training Week 4 | 219.63 (67.55) | 225.35 (75.05)

5. Secondary Outcome: Mean Motor Activity Log (MAL) Score: Amount Subtest
Description: Individuals are asked to rate amount of movement during 30 daily functional tasks. Items are scored on a 0 to 6-point ordinal scale as follows:
  0 = The weaker arm was not used at all for that activity (never)
  1 = Occasionally used weaker arm, but only very rarely (very rarely)
  2= Sometimes used weaker arm, but did the activity most of the time with stronger arm (rarely)
  3 = Used weaker arm about half as much as before the stroke (half pre-stroke)
  4 = Used weaker arm almost as much as before the stroke (3/4 pre-stroke)
  5 = The ability to use the weaker arm for that activity was as good as before the stroke (normal)
  Total scores range from 0 to 140; 0 indicating the least movement 140 indicating the most movement. The scores were converted into percentage scores where higher percent score indicate more movement and lower percent score less movement.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 78.67 (23.16) | 78.00 (24.76)
  Post-Training Week 1 | 81.00 (23.63) | 79.00 (25.39)
  Post-Training Week 4 | 84.67 (23.21) | 77.33 (25.42)

6. Secondary Outcome: Mean Motor Activity Log (MAL): How Well Subtest
Description: Individuals are asked to rate quality of movement during 30 daily functional tasks. Items are scored on a 6-point ordinal scale as follows:
  0=The weaker arm was not used at all for that activity (never); 1=The weaker arm was moved during that activity, but was not helpful (very poor); 2=The weaker arm was of some use during the activity, but needed help from the stronger arm or moved very slowly or with difficulty (poor); 3=The weaker arm was used for the purpose indicated, but movements were slow or were made with only some effort (fair); 4=The movements made by the weaker arm were almost normal, but were not quite as fast or accurate as normal (almost normal); 5=The ability to use the weaker arm for that activity was as good as before the stroke (normal)
  Total scores range from 0 to 140; 0 indicating the least movement and 140 indicating the most movement.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 3.41 (.96) | 3.17 (1.18)
  Post-Training Week 1 | 3.64 (1.04) | 3.48 (1.23)
  Post-Training Week 4 | 3.92 (.96) | 3.33 (1.21)

7. Secondary Outcome: Mean Wolf Motor Function Test (WMFT) Total Time
Description: The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks. There are 15 timed tasks included with a time cap of 120 seconds. The max amount of time to completion is 1800 seconds if all tasks are failed. The time in seconds were summed across all the tasks to obtain the total duration. Values in the table represent the time taken in seconds to successfully complete all 15 tasks).
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 120.84 (230.77) | 130.04 (153.06)
  Post-Training Week 1 | 91.31 (169.83) | 99.02 (131.79)
  Post-Training Week 4 | 99.81 (206.77) | 91.42 (118.77)

8. Secondary Outcome: Mean Wolf Motor Function Test Functional Ability (WMFT-FS) Scale Score
Description: The WMFT is a 17 item scale that quantifies upper extremity (UE) motor ability through timed and functional tasks. The items are rated on a 6-point scale.Total scores can range from 17 to 102. Lower scores indicate debilitating mobility (such as no or limited functionality), while higher score indicate greater mobility (such as slow movement and normal movement).
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: One participant from both arms was removed from the data analysis due to errors in data collection yielding uninterpretable results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 4.07 (.57) | 4.08 (.72)
  Post-Training Week 1 | 4.31 (.55) | 4.29 (.62)
  Post-Training Week 4 | 4.34 (.54) | 4.13 (.54)

9. Secondary Outcome: Mean Wolf Motor Function Test (WMFT) Grip Strength
Description: Participants attempt to grip the dynamometer with greatest grip strength possible. The test should be conducted 3 times with a 1-minute rest between trials. The mean of grip strength exerted (kg) on 3 trials is then calculated.
Time Frame: Baseline, Post-Training (1 Week), Post-Training (4 Weeks)
Population: Analysis was conducted for participants that completed all study procedures.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Number analyzed (Participants) | 10 | 10
kilograms
  Baseline | 20.80 (13.98) | 22.30 (12.72)
  Post-Training Week 1 | 22.30 (19.10) | 20.30 (9.04)
  Post-Training Week 4 | 20.90 (13.73) | 20.00 (11.57)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline measurements through week 5.
Arm/Group | Hebbian-type Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes